CLINICAL TRIAL: NCT01776593
Title: The Best Parameter of Bladder Diary Correlates With the Volume at Strong Desire to Void of Filling Cystometry
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Professor, Ho-Hsiung Lin, National Taiwan University Hospital
Other Study IDs: 201203078RIC
Record Dates: First submitted 2013-01-18; First posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Bladder Diary; Urodynamic Studies
Keywords: bladder capacity; bladder diary; bladder oversensitivity; lower urinary tract symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lower urinary tract symptoms

SUMMARY:
To identify the bladder diary parameters that are best correlated to VSD.

DETAILED DESCRIPTION:
To identify the bladder diary parameters that are best correlated to VSD.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with lower urinary tract symptoms who had underwent urodynamic studies

Exclusion Criteria:

* Patients without data of bladder diary

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with lower urinary tract symptoms
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To identify the bladder diary parameter that is best correlated to the volume at strong desire to void of filling cystometry. | 1 week
  To identify which bladder diary parameter that is best correlated to the volume at strong desire to void of filling cystometry. Thus, that bladder diary parameter may be used as a surrogate for the volume of strong desire to void of filling cystometry and without the need of urodynamic studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics & Gynecology, National Taiwan University Hospital, Taipei, Taiwan, Taiwan